CLINICAL TRIAL: NCT02068040
Title: Effects of Epicatechin on Functional Capacity, Skeletal Muscle Structure and Diastolic Function in Patients With Heart Failure With Preserved Ejection Fraction (HFPEF)
Acronym: HFPEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Pam Taub, MD, Dr. Pam Taub, University of California, San Diego
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD IRB 130398
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure
Keywords: with preserved ejection fraction of >55%
MeSH Terms: conditions — Heart Failure

ARMS (1):
- CocoaVia capsules (Experimental): From baseline to 3 months, patients will consume 2 capsules containing pure epicatechin
  Interventions: Dietary Supplement: CocoaVia

INTERVENTIONS:
Dietary Supplement: CocoaVia — CocoaVia contains flavanols found natrually in cocoa beans. Capsules will contain 250mg of flavanol
  Other Names: Epicatechin consumption

SUMMARY:
The major goal of this proposal is to characterize the ability of epicatechin which a component of dark chocolate to improve the

1. structural and functional features of skeletal muscle (SkM)
2. exercise capacity (as assessed by VO2 max)
3. parameters of diastolic heart function (as assessed by echocardiography)

We propose that a 3 month treatment with epicatechin (through CocoaVia® capsules) will lead to a significant improvement in exercise capacity and diastolic function.

DETAILED DESCRIPTION:
Patient Inclusion/Exclusion Criteria:

1. New York Heart Association Class II/III HF with preserved ejection fraction (EF) of >50%.
2. Nonsmokers
3. Subject not taking Coumadin, Xarelto, Prasugrel or Pradaxa. Patients on Plavix for drug eluting stent will not be excluded.
4. Ages between 40-65. We will exclude any women of child bearing potential

ELIGIBILITY:
Inclusion Criteria:

* Medically Diagnosed Heart Failure with Ejection Fraction of >55%
* BMI 27-32
* No Significant HbA1C fluctuations in past 6 months

Exclusion Criteria:

* Smoking or quit smoking less than 1 year prior to enrollment
* Substance Abuse
* Taking Coudmadin or Pradaxa

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in exercise capacity | Baseline and 3 months
  Objectively evaluate exercise capacity through cycle ergometry to measure VO2 max
Change from baseline in skeletal muscle metabolism | Baseline and 3 months
  The change in skeletal muscle metabolism will be evaluated by magnetic resonance spectroscopy
Change from baseline in pre-specified biomarker levels in blood, skeletal muscle, and urine | Baseline and 3 months
  Skeletal muscle biopsies and blood draws will be performed to obtain experimental samples

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Taub PR, Ramirez-Sanchez I, Ciaraldi TP, Perkins G, Murphy AN, Naviaux R, Hogan M, Maisel AS, Henry RR, Ceballos G, Villarreal F. Alterations in skeletal muscle indicators of mitochondrial structure and biogenesis in patients with type 2 diabetes and heart failure: effects of epicatechin rich cocoa. Clin Transl Sci. 2012 Feb;5(1):43-7. doi: 10.1111/j.1752-8062.2011.00357.x. Epub 2011 Nov 7. PMID 22376256